CLINICAL TRIAL: NCT02509507
Title: A Phase 1b/2, Multicenter, Open-label, Basket Trial to Evaluate the Safety of Talimogene Laherparepvec Injected Into Liver Tumors Alone and in Combination With Systemic Pembrolizumab in Phase 1b and to Evaluate the Efficacy and Safety of Intratumoral Talimogene Laherparepvec in Combination With Systemic Pembrolizumab to Treat Subjects With Advanced Solid Tumors in Phase 2 (MASTERKEY-318)
Brief Title: Trial to Evaluate the Safety of Talimogene Laherparepvec Injected Into Tumors Alone and in Combination With Systemic Pembrolizumab MK-3475-611/Keynote-611
Acronym: MASTERKEY-318
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20140318; 2014-005386-67 (EudraCT Number)
Record Dates: First submitted 2015-07-10; First posted 2015-07-28 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma; Liver Metastases; Cutaneous or Subcutaneous Lymph Node; Liver Tumors
Keywords: Liver tumours
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — talimogene laherparepvec; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase Ib/II Talimogene Laherparepvec (Experimental): Talimogene Laherparepvec
  Interventions: Drug: Talimogene Laherparepvec
- Phase Ib/II Talimogene Laherparepvec + Pembrolizumab (Experimental): Combination treatment of Talimogene Laherparepvec and Pembrolizumab
  Interventions: Drug: Talimogene Laherparepvec; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene laherparepvec (T-VEC) administered by intralesional injection into liver tumors, with ultrasound/computed tomography (US/CT) guidance. Part 1: initial dose of T-VEC is 10^6 plaque forming unit (PFU)/mL up to 4mL in Cohorts 1 & 2, up to 8mL in Cohorts 3 & 4 of the Group A & Group B. The 1st cycle of T-VEC will be 21 (+3) days (from the 1st dose at 10^6 PFU/mL to the 2nd dose at 10^7 or 10^8 PFU/mL). Subsequent cycles of T-VEC will be 21 (±3) days. Max. volume of T-VEC administered at any dose is 4mL (Cohorts 1, 2, 5, and 6) or 8mL (Cohorts 3 & 4) for any individual lesion or for all lesions combined. Part 2: Initial dose of T-VEC is 10^6 PFU/mL followed by subsequent T-VEC doses at a concentration of 10^8 PFU/mL. T-VEC volume is up to 8mL based on the size of the inejected lesions. NOTE: as of Protocol Amendment 6 [dated 26 October 2021], intrahepatic injections of talimogene laherparepvec and liver biopsies are no longer performed in this study.
Drug: Pembrolizumab — Pembrolizumab is a non-Amgen Investigational product that is manufactured by Merck. Pembrolizumab will be labeled, packaged, and distributed by Amgen (or designee) using Amgen (or designee) clinical study drug distribution procedures. Pembrolizumab is supplied as pembrolizumab 100 mg/4 mL vials (25 mg/mL) solution for IV infusion. The trial treatment will consist of a total dose of 200mg administered intravenously every 3 weeks (day 1 of each cycle) for up to 35 cycles.
  Arms: Phase Ib/II Talimogene Laherparepvec + Pembrolizumab

SUMMARY:
This is a phase 1b/2, multicenter, open-label, basket trial to evaluate the safety of talimogene laherparepvec injected intrahepatically into liver tumors alone and in combination with systemic intravenous (IV) administration of pembrolizumab, in subjects with non-hepatocellular carcinoma (HCC) liver metastases from breast adenocarcinoma (BC), colorectal adenocarcinoma (CRC), gastroesophageal cancer (GEC), melanoma, non-small cell lung cancer (NSCLC), clear cell renal cell carcinoma (RCC) in Part 1 Group A, and subjects with HCC with and without viral hepatitis in Part 1 Group B (viral hepatitis is only applicable in combination setting), and to evaluate the efficacy and safety of intratumoral talimogene laherparepvec in combination with systemic pembrolizumab in subjects with advanced triple negative breast cancer (TNBC), hormone receptor positive breast cancer, CRC, cutaneous squamous cell carcinoma (CSCC), and basal cell carcinoma (BCC) in Part 2 Group A and subjects with HCC with and without viral hepatitis in Part 2 Group B. The objective of Part 1 is to evaluate the safety of intrahepatic injection of talimogene laherparepvec into liver tumors alone and in combination with systemically administered pembrolizumab for the non-HCC (Group A) and HCC (Group B) cohorts separately. Part 2 consists of 2-stage design to evaluate the efficacy and safety of talimogene laherparepvec in combination with systemic pembrolizumab. Efficacy and safety will be evaluated in each of the five non-HCC tumor types from Group A separately. Similarly, the efficacy and safety of the combination treatment will be determined for Group B HCC subjects. As of Protocol Amendment 6 (dated 26 October 2021), intrahepatic injections of talimogene laherparepvec and liver biopsies are no longer performed in this study. Enrollment for this study has stopped.

ELIGIBILITY:
Summary of Subject Eligibility Criteria:

Key Inclusion Criteria:

Subjects must be age ≥ 18 years at the time of informed consent. Subjects must have histologically or cytologically confirmed disease.

Part 1 is restricted to BC, CRC, GEC, melanoma, NSCLC, or RCC with liver metastases or HCC.

Part 2 Group A is restricted to advanced hormone receptor positive BC, CRC, TNBC, CSCC, and BCC with or without liver metastases.

* Part 2 Hormone receptor positive Breast Cancer Arm only: Histologically and/or cytologically confirmed diagnosis of estrogen receptor (ER) positive and/or progesterone receptor (PrR) positive breast cancer.
* Triple negative breast cancer: Histologically and/or cytologically confirmed diagnosis of ER negative, PrR negative, human epidermal growth factor receptor 2 (HER2)-Neu negative.

Part 2 Group B is restricted to HCC (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible).

For HCC subjects with a diagnosis of hepatitis B, they must be on antiviral therapy for at least 4 weeks prior to enrollment and hepatitis B virus (HBV) viral load by real-time polymerase chain reaction (qPCR) must be < 100 IU/mL. HCC subjects with past or ongoing hepatitis C infection must have completed treatment for hepatitis C at least 1 month prior to study enrollment and hepatitis C viral load must be undetectable; subjects with hepatitis B and C must fulfill the eligibility criteria for hepatitis B and hepatitis C. Subjects with unresectable locally recurrent TNBC are eligible.

Non-HCC subjects must have received at least 1 prior standard of care systemic anti-cancer therapy for their locally advanced or metastatic disease. For the combination cohorts (Cohorts 5 and 6 in Part 1) and Part 2, subjects with melanoma CSCC or NSCLC do not need to have received prior therapy. In Part 1, subjects must have measurable liver tumors and liver tumors that are suitable for injection. In Part 2, subjects must have measurable disease and cutaneous, subcutaneous, lymph node, or liver tumors suitable for injection. NOTE: as of Protocol Amendment 6 [dated 26 October 2021], intrahepatic injections of talimogene laherparepvec and liver biopsies are no longer performed in this study, enrollment for this study has stopped. Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1, and life expectancy should be approximately 5 months or more. Adequate hematological, renal, hepatic, and coagulation function is required. Liver function tests may be mildly abnormal but within the parameters. Child-Pugh score must be A.

Key Exclusion Criteria:

Subjects must not be candidates for surgery or locoregional therapy with curative intent or planned systemic anti-cancer therapy, with the exception of immunotherapy in the combination cohorts (Cohorts 5 and 6 in Part 1 and all subjects in Part 2). Liver tumors must not be estimated to invade approximately more than one-third of the liver. Liver tumor-directed therapy, hepatic surgery or major surgery, antibody-based therapy, or immunotherapy must not have been performed < 28 days, chemotherapy < 21 days, and targeted small molecule therapy or hormonal therapy < 14 days prior to enrollment. Subjects must either (1) have no central nervous system (CNS) metastasis, or carcinomatous meningitis, or (2) if CNS metastasis is present, must have stable treated cerebral metastases. Subjects must not have symptomatic auto-immune disease or be symptomatically immunosuppressed. They must not have a history of solid organ transplantation. For non-HCC, there must not be acute or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. For HCC with prior hepatitis B and/or C infection, HBV and/or HCV viral load by qPCR must be undetectable, and they must not have had recent treatment within 12 weeks for HBV or HCV with certain antiviral medications in Part 1 Group B cohorts 1-5 and 6a, and Part 2 Group B HCC without viral hepatitis. For all patients in Part 1 and for patients in Part 2 where intrahepatic liver injection is planned (NOTE: as of Protocol Amendment 6 [dated 26 October 2021], intrahepatic injections of talimogene laherparepvec and liver biopsies are no longer performed in this study, enrollment for this study has stopped), there should be no macroscopic intravascular invasion of tumors into the main portal vein, hepatic vein, or vena cava. Subjects must not: have active herpetic skin lesions or prior complications of herpetic infection (eg, herpetic keratitis or encephalitis); require treatment with an antiherpetic drug; have received live-virus vaccination within 30 days of planned treatment start; have previous therapy with talimogene laherparepvec, oncolytic viruses, or tumor vaccine. Subjects in the combination treatment cohort must not have: a history or evidence of psychiatric, substance abuse, or any other clinically significant disorder; toxic effects of the most recent prior chemotherapy not resolved to grade 1 or less (except alopecia); or expected other cancer therapy while on study with the exception of local radiation to the site of bone or other metastasis for palliative treatment. Male subjects of reproductive potential in the combination treatment must be willing to use acceptable methods of effective contraception during treatment and through 4 months after the last dose of pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (32):
- United States (9):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California Los Angeles, Santa Monica, California
  - Georgetown-Howard University Center for Clinical Translational Science, Washington D.C., District of Columbia
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Washington University School of Medicine, Center for Advanced Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Tasman Oncology Research, Southport, Queensland
- Landeskrankenhaus Salzburg, Salzburg, Austria
- Belgium (3):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- Germany (4):
  - Charite Universitätsmedizin Berlin, Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Kreiskliniken Reutlingen - Klinikum am Steinenberg, Reutlingen
  - Universitätsklinikum Tübingen, Tübingen
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- South Korea (3):
  - Cha Bundang Medical Center, Cha University, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (4):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Switzerland (4):
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Winterthur, Winterthur
  - Universitaetsspital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Hecht JR, Oberoi A, Garralda Cabanas E, Jae Chon H, Digklia A, Rottey S, Martin Jimenez M, Chaney M, Hippenmeyer J, Lawrence T, Liu K, Hamidi A, Chesney J. Phase Ib/II trial of talimogene laherparepvec alone and with pembrolizumab in advanced solid tumors with liver metastases and hepatocellular carcinoma. Oncologist. 2025 Mar 10;30(3):oyae203. doi: 10.1093/oncolo/oyae203. PMID 40156118
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 127 participants were enrolled at 22 centers in Australia, Europe, South Korea and the United States from February 2016 to July 2023.
  As of protocol amendment 6 (dated 26 October 2021), intrahepatic injections of talimogene laherparepvec were no longer performed.
Pre-assignment Details: Of the 190 participants screened, 127 participants were enrolled and received study treatment.
Groups:
- Part 1: Monotherapy Group A: Participants with non-hepatocellular carcinoma (non-HCC) were administered talimogene laherparepvec by intralesional injection at an initial concentration of 10^6 plaque forming unit (PFU)/mL in a volume of up to 4mL in Cohorts 1 & 2 and up to a volume of 8 mL in Cohorts 3 & 4 on Day 1 of the first 21-day cycle. The concentration of talimogene laherparepvec doses in the second and subsequent 21-day cycles were 10^7 (Cohorts 1 & 4) or 10^8 PFU/mL (Cohorts 2 & 3).
- Part 1: Monotherapy Group B: Participants with hepatocellular carcinoma (HCC) were administered talimogene laherparepvec by intralesional injection at an initial concentration of 10^6 plaque forming unit (PFU)/mL in a volume of up to 4mL in Cohorts 1 & 2 and up to a volume of 8 mL in Cohorts 3 & 4 on Day 1 of the first 21-day cycle. The concentration of talimogene laherparepvec doses in the second and subsequent 21-day cycles were 10^7 (Cohorts 1 & 4) or 10^8 PFU/mL (Cohorts 2 & 3).
- Part 1: Combination Therapy Group A: Participants with non-hepatocellular carcinoma (non-HCC) were administered talimogene laherparepvec by intralesional injection at an initial concentration of 10^6 plaque forming unit (PFU)/mL in a volume of up to 4mL in Cohorts 5 & 6 on Day 1 of the first 21-day cycle. The concentration of talimogene laherparepvec doses in the second and subsequent 21-day cycles were 10^7 (Cohort 5) or 10^8 PFU/mL (Cohorts 6).
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
- Part 1: Combination Therapy Group B: Participants with hepatocellular carcinoma (HCC) were administered talimogene laherparepvec by intralesional injection at an initial concentration of 10^6 plaque forming unit (PFU)/mL in a volume of up to 4mL in Cohorts 5, 6a (participants without viral hepatitis) and 6b (participants with well controlled viral hepatitis) on Day 1 of the first 21-day cycle. The concentration of talimogene laherparepvec doses in the second and subsequent 21-day cycles were 10^7 (Cohort 5) or 10^8 PFU/mL (Cohorts 6a and 6b).
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
- Part 2: Hormone Receptor Positive Breast Cancer (HRBC): Participants with HRBC were administered talimogene laherparepvec by intralesional injection at the maximum tolerated concentration (MTC) and maximum tolerated volume (MTV) identified in Part 1 on Day 1 of each 21-day cycle.
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
- Part 2: Triple Negative Breast Cancer (TNBC): Participants with TNBC were administered talimogene laherparepvec by intralesional injection at the MTC and MTV identified in Part 1 on Day 1 of each 21-day cycle.
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
- Part 2: Cutaneous Squamous Cell Carcinoma (CSCC): Participants with CSCC were administered talimogene laherparepvec by intralesional injection at the MTC and MTV identified in Part 1 on Day 1 of each 21-day cycle.
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
- Part 2: Basal Cell Carcinoma (BCC): Participants with BCC were administered talimogene laherparepvec by intralesional injection at the MTC and MTV identified in Part 1 on Day 1 of each 21-day cycle.
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
- Part 2: Colorectal Adenocarcinoma (CRC): Participants with CRC were administered talimogene laherparepvec by intralesional injection at the MTC and MTV identified in Part 1 on Day 1 of each 21-day cycle.
  Participants were also administered 200 mg of pembrolizumab on Day 1 of each 21-day cycle as an intravenous infusion.
Period: Overall Study
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Started | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
Received Talimogene Laherparepvec | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
Received Pembrolizumab | 0 | 0 | 24 | 22 | 10 | 18 | 10 | 5 | 10
Completed | 0 | 1 | 1 | 4 | 1 | 1 | 1 | 1 | 1
Not Completed | 23 | 4 | 23 | 18 | 9 | 17 | 9 | 4 | 9
Not completed — Death | 21 | 3 | 22 | 14 | 8 | 12 | 5 | 4 | 8
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 4 | 1 | 3 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Part 1 - Included all participants who have received at least 1 dose of talimogene laherparepvec in monotherapy arms, and at least 1 dose of talimogene laherparepvec or at least 1 dose of pembrolizumab in combination arms. Part 2 - Included all participants who have received at least 1 dose of talimogene laherparepvec or at least 1 dose of pembrolizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC) | Total
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10 | 127
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 16 | 3 | 17 | 10 | 8 | 15 | 5 | 4 | 6 | 84
  65 - 74 years | 7 | 2 | 5 | 8 | 2 | 2 | 2 | 1 | 4 | 33
  75 - 84 years | 0 | 0 | 2 | 4 | 0 | 1 | 3 | 0 | 0 | 10
  >= 85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 10 | 5 | 10 | 18 | 3 | 2 | 4 | 65
  Male | 12 | 3 | 14 | 17 | 0 | 0 | 7 | 3 | 6 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 8
  Not Hispanic or Latino | 21 | 5 | 23 | 21 | 10 | 16 | 9 | 4 | 10 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 8 | 0 | 3 | 3 | 1 | 1 | 19
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 20 | 4 | 23 | 14 | 10 | 15 | 7 | 4 | 9 | 106
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: All toxicities were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03:
  * Grade 1: Mild
  * Grade 2: Moderate
  * Grade 3: Severe or medically significant but not immediately life threatening
  * Grade 4: Life threatening consequences
  * Grade 5: Death related to adverse event (AE)
  The occurrence of specific pre-defined toxicities during the DLT evaluation period were considered a DLT if judged by the investigator to be related to talimogene laherparepvec and/or pembrolizumab.
  All Grade 5 toxicities, intolerable toxicities that lead to permanent discontinuation of talimogene laherparepvec and/or pembrolizumab and Grade 3 or higher AEs related to talimogene laherparepvec and/or pembrolizumab that resulted in a study treatment delay by > 2 weeks were considered DLTs.
Time Frame: Cycle 1 and Cycle 2: Day 1 to Day 21
Population: DLT Analysis Set: Participants who had at least 1 dose of planned monotherapy or combination treatment and had the opportunity to be on treatment for at least 6 weeks from the initial dosing of study treatment & received at least 1 additional dose of monotherapy or combination or experienced a DLT during the DLT-evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 18 | 5 | 20 | 19 | 8 | 11 | 5 | 4 | 9
Participants | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2 Only: Objective Response Rate (ORR) Per Modified Immune-related Response Criteria Simulating Response Evaluation Criteria in Solid Tumors (irRC-RECIST).
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) per modified irRC-RECIST.
  * CR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
Time Frame: Up to 154 weeks
Population: Full Analysis Set (Part 2): Included all participants in Part 2 who received at least 1 dose of talimogene laherparepvec and at least 1 dose of pembrolizumab in combination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 10 | 18 | 10 | 5 | 10
percentage of participants | 10.0 [0.3 to 44.5] | 16.7 [3.6 to 41.4] | 10.0 [0.3 to 44.5] | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 30.8]

3. Primary Outcome: Part 2 Only: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an event that emerged during treatment, having been absent pretreatment, or worsened relative to the pretreatment state.
  A treatment-related TEAE was defined as a TEAE that was suspected to be related to the study treatment.
Time Frame: Day 1 to 30 days post-last dose of talimogene laherparepvec or pembrolizumab, whichever is later. The maximum duration of talimogene laherparepvec treatment was 102.4 weeks and pembrolizumab treatment was 109.3 weeks in Part 2.
Population: Safety Analysis Set (Part 2): Included all participants in Part 2 who have received at least 1 dose of talimogene laherparepvec or at least 1 dose of pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 10 | 18 | 10 | 5 | 10
Participants
  TEAEs | 10 | 17 | 9 | 5 | 10
  Treatment-related TEAEs | 10 | 12 | 4 | 5 | 10

4. Secondary Outcome: Part 1 Only: ORR Per Modified irRC-RECIST
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR per modified irRC-RECIST.
  * CR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
Time Frame: Up to 297 weeks
Population: Full Analysis Set (Part 1): Included all participants in Part 1 who received at least 1 dose of talimogene laherparepvec in monotherapy and combination cohorts and at least 1 dose of pembrolizumab in combination cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B
Number analyzed (Participants) | 23 | 5 | 24 | 22
percentage of participants | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 52.2] | 8.3 [1.0 to 27.0] | 13.6 [2.9 to 34.9]

5. Secondary Outcome: Best Overall Response (BOR) Per Modified irRC-RECIST
Description: BOR was defined as the number of participants with a best visit response in the following order: CR, PR, stable disease (SD), progressive disease (PD), or unevaluable (UE) as per modified irRC-RECIST.
  * CR: Disappearance of all lesions and confirmation by assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
  * SD: Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.
  * PD: Increase in tumor burden ≥ 20 % and at least 5 mm absolute increase relative to nadir confirmation by a repeat, consecutive assessment no less than 4 weeks (28 days) from the date first documented PD.
  * UE: Any lesion present at baseline which was not assessed or was unable to be evaluated.
Time Frame: Up to 297 weeks
Population: Full Analysis Set: Included all participants who received at least 1 dose of talimogene laherparepvec in monotherapy and combination cohorts and at least 1 dose of pembrolizumab in combination cohorts in Part 1 and Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  PR | 0 | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 0
  SD | 1 | 1 | 4 | 6 | 1 | 1 | 1 | 2 | 3
  PD | 7 | 1 | 10 | 3 | 3 | 5 | 2 | 0 | 1
  UE | 13 | 3 | 7 | 10 | 5 | 6 | 4 | 2 | 5
  Not Done | 2 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 1

6. Secondary Outcome: Durable Response Rate (DRR) Per Modified irRC-RECIST
Description: DRR per modified irRC-RECIST was defined as the percentage of participants with an objective response (CR/PR) with a duration of response of at least 6 months.
  * CR: Disappearance of all lesions and confirmation by assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
Time Frame: Up to 297 weeks
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
percentage of participants | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 52.2] | 8.3 [1.0 to 27.0] | 9.1 [1.1 to 29.2] | 10.0 [0.3 to 44.5] | 11.1 [1.4 to 34.7] | 10.0 [0.3 to 44.5] | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 30.8]

7. Secondary Outcome: Duration of Response (DOR) Per Modified irRC-RECIST
Description: DOR per modified irRC-RECIST was defined as the time from the date of an initial response (CR/PR) that was subsequently confirmed to the earlier of PD or death. DOR was estimated using the Kaplan-Meier method.
  * CR: Disappearance of all lesions and confirmation by assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
  * PD: Increase in tumor burden ≥ 20 % and at least 5 mm absolute increase relative to nadir confirmation by a repeat, consecutive assessment no less than 4 weeks (28 days) from the date first documented PD.
Time Frame: Up to 297 weeks
Population: Full Analysis Set: Included all participants who received at least 1 dose of talimogene laherparepvec in monotherapy and combination cohorts and at least 1 dose of pembrolizumab in combination cohorts in Part 1 and Part 2. Only participants who had a BOR of CR/PR were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3 | 1 | 1 | 0
months |  |  | 16.8 [12.2 to NA] — Due to limited number of events, upper limit was not reached. | 8.9 [4.3 to NA] — Due to limited number of events, upper limit was not reached. | NA [NA to NA] — Due to limited number of events, median and upper/lower limits were not reached. | 23.1 [5.1 to NA] — Due to limited number of events, upper limit was not reached. | NA [NA to NA] — Due to limited number of events, median and upper/lower limits were not reached. | NA [NA to NA] — Due to limited number of events, median and upper/lower limits were not reached. |

8. Secondary Outcome: Disease Control Rate (DCR) Per Modified irRC-RECIST
Description: DCR per modified irRC-RECIST was defined as percentage of participants that had a BOR in 1 of the following: CR, PR or SD.
  * CR: Disappearance of all lesions and confirmation by assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
  * SD: Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.
Time Frame: Up to 297 weeks
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
percentage of participants | 4.3 [0.1 to 21.9] | 20.0 [0.5 to 71.6] | 25.0 [9.8 to 46.7] | 40.9 [20.7 to 63.6] | 20.0 [2.5 to 55.6] | 22.2 [6.4 to 47.6] | 20.0 [2.5 to 55.6] | 60.0 [14.7 to 94.7] | 30.0 [6.7 to 65.2]

9. Secondary Outcome: Progression Free Survival (PFS) Per Modified irRC-RECIST
Description: PFS was defined as the time from first dose to the date of first of PD per modified irRC-RECIST criteria, or death, whichever occurs first. PFS was estimated using the Kaplan-Meier method. Participants that did not have an event of death or disease progression were censored at the latter of their last evaluable tumor assessment date or first dose date.
  * PD: Increase in tumor burden ≥ 20 % and at least 5 mm absolute increase relative to nadir confirmation by a repeat, consecutive assessment no less than 4 weeks (28 days) from the date first documented PD.
Time Frame: Up to 297 weeks
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
months | 2.3 [1.9 to 9.0] | 3.9 [1.9 to NA] — Due to limited number of events, data were not evaluable. | 2.0 [1.9 to 6.2] | 8.1 [3.2 to 13.2] | 6.1 [1.6 to 20.5] | 2.9 [1.2 to 10.2] | 5.4 [2.2 to NA] — Due to limited number of events, data were not evaluable. | 16.4 [5.4 to NA] — Due to limited number of events, data were not evaluable. | 8.8 [2.4 to 12.5]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose date to the date of death from any cause. OS time was censored at the last date the participant was known to be alive when the confirmation of death was absent or unknown, or at the date 24 months after the last participant enrolled if the last known to be alive/death date was beyond it. One month = 365.25/12 days. OS was estimated using the Kaplan-Meier method.
Time Frame: Up to 297 weeks
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
months | 8.7 [2.7 to 17.1] | 9.1 [3.9 to NA] — Due to limited number of events, upper limit was not reached. | 7.8 [4.4 to 14.2] | 12.8 [6.8 to 29.5] | 9.1 [2.4 to 20.5] | 10.2 [2.7 to 27.2] | 9.6 [2.3 to NA] — Due to limited number of events, upper limit was not reached. | 16.4 [5.4 to NA] — Due to limited number of events, upper limit was not reached. | 11.2 [2.4 to 18.9]

11. Secondary Outcome: Part 1 Only: Number of Participants Who Experienced a TEAE
Description: as for outcome 3
Time Frame: Day 1 to 30 days post-last dose of talimogene laherparepvec or pembrolizumab, whichever is later. The maximum duration of talimogene laherparepvec treatment was 34.1 weeks and pembrolizumab treatment was 98.3 weeks in Part 1.
Population: Safety Analysis Set (Part 1): Included all participants in Part 1 who have received at least 1 dose of talimogene laherparepvec or at least 1 dose of pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B
Number analyzed (Participants) | 23 | 5 | 24 | 22
Participants
  TEAEs | 23 | 5 | 24 | 21
  Treatment-related TEAEs | 23 | 5 | 22 | 20

12. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Deoxyribonucleic Acid (DNA) in Blood
Description: Blood samples were tested using real-time polymerase chain reaction (qPCR). Detectable DNA was defined as a positive result by qPCR analysis.
Time Frame: Week 1 to Week 10
Population: Blood Evaluable Analysis Set: Included all participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one post dose blood sample collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
percentage of participants | 100.0 [85.2 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [85.8 to 100.0] | 95.5 [77.2 to 99.9] | 90.0 [55.5 to 99.7] | 88.9 [65.3 to 98.6] | 50.0 [18.7 to 81.3] | 60.0 [14.7 to 94.7] | 100.0 [69.2 to 100.0]

13. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA in Urine
Description: Urine samples were tested using qPCR. Detectable DNA was defined as a positive result by qPCR analysis.
Time Frame: Week 1 to Week 10
Population: Urine Evaluable Analysis Set: Included all participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one post dose urine sample collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 18 | 10 | 5 | 10
percentage of participants | 34.8 [16.4 to 57.3] | 40.0 [5.3 to 85.3] | 37.5 [18.8 to 59.4] | 54.5 [32.2 to 75.6] | 10.0 [0.3 to 44.5] | 27.8 [9.7 to 53.5] | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 52.2] | 30.0 [6.7 to 65.2]

14. Secondary Outcome: Percentage of Participants With Clearance of Talimogene Laherparepvec in Blood
Description: Blood samples were tested using qPCR.
  A participant was defined as having cleared talimogene laherparepvec if a negative qPCR in a sample was obtained following a prior positive test and if there were no subsequent positive test results in the same cycle.
Time Frame: Cycles 2, 3 and 4: Day 1 pre-dose. Each cycle was 21 days.
Population: Blood Clearance Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least 2 post dose samples, collected within the same dosing cycle. Participants must have had at least 1 positive sample and at least 1 subsequent sample at any time during the cycle. All participants included in the overall number of participants contributed analyzed data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 21 | 9 | 16 | 5 | 3 | 10
percentage of participants
  Cycle 2, Day 1 Pre-dose: number analyzed (Participants) | 23 | 5 | 23 | 21 | 7 | 15 | 3 | 3 | 10
  Cycle 2, Day 1 Pre-dose | 73.9 [51.6 to 89.8] | 100.0 [47.8 to 100.0] | 52.2 [30.6 to 73.2] | 95.2 [76.2 to 99.9] | 85.7 [42.1 to 99.6] | 80.0 [51.9 to 95.7] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 60.0 [26.2 to 87.8]
  Cycle 3, Day 1 Pre-dose: number analyzed (Participants) | 18 | 5 | 20 | 18 | 9 | 12 | 4 | 2 | 10
  Cycle 3, Day 1 Pre-dose | 66.7 [41.0 to 86.7] | 100.0 [47.8 to 100.0] | 70.0 [45.7 to 88.1] | 100.0 [81.5 to 100.0] | 77.8 [40.0 to 97.2] | 75.0 [42.8 to 94.5] | 75.0 [19.4 to 99.4] | 100.0 [15.8 to 100.0] | 70.0 [34.8 to 93.3]
  Cycle 4, Day 1 Pre-dose: number analyzed (Participants) | 3 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4, Day 1 Pre-dose | 66.7 [9.4 to 99.2] |  | 37.5 [8.5 to 75.5] |  |  |  |  |  | 100.0 [2.5 to 100.0]

15. Secondary Outcome: Percentage of Participants With Clearance of Talimogene Laherparepvec in Urine
Description: Urine samples were tested using qPCR.
  A participant was defined as having cleared talimogene laherparepvec if a negative qPCR in a sample was obtained following a prior positive test and if there were no subsequent positive test results in the same cycle.
Time Frame: Cycles 2, 3 and 4: Day 1 pre-dose. Each cycle was 21 days.
Population: Urine Clearance Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least 2 post dose samples, collected within the same dosing cycle. Participants must have had at least 1 positive sample and at least 1 subsequent sample at any time during the cycle. All participants included in the overall number of participants contributed analyzed data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 8 | 2 | 9 | 11 | 1 | 5 | 1 | 0 | 3
percentage of participants
  Cycle 2, Day 1 Pre-dose: number analyzed (Participants) | 3 | 1 | 5 | 3 | 0 | 3 | 1 | 0 | 2
  Cycle 2, Day 1 Pre-dose | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [29.2 to 100.0] |  | 100.0 [29.2 to 100.0] | 0.0 [0.0 to 97.5] |  | 100.0 [15.8 to 100.0]
  Cycle 3, Day 1 Pre-dose: number analyzed (Participants) | 7 | 1 | 5 | 10 | 1 | 3 | 0 | 0 | 2
  Cycle 3, Day 1 Pre-dose | 100.0 [59.0 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] |  |  | 100.0 [15.8 to 100.0]
  Cycle 4, Day 1 Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA at the Surface of Injection Site
Description: The number of participants with positive qPCR and subsequent positive plaque assays were evaluated from swabs of skin surface of injections. Detectable DNA was defined as a positive result by qPCR analysis.
Time Frame: Week 1 to Week 10
Population: Skin Surface of Injections Evaluable Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the skin surface of injections.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 16 | 10 | 4 | 10
percentage of participants | 69.6 [47.1 to 86.8] | 60.0 [14.7 to 94.7] | 79.2 [57.8 to 92.9] | 72.7 [49.8 to 89.3] | 60.0 [26.2 to 87.8] | 68.8 [41.3 to 89.0] | 80.0 [44.4 to 97.5] | 100.0 [39.8 to 100.0] | 60.0 [26.2 to 87.8]

17. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus at the Surface of Injection Site
Description: The percentage of participants with detectable virus were evaluated from swabs of skin surface of injections. Detectable virus was defined as a positive result by TCID50.
Time Frame: Week 1 to Week 10
Population: Skin Surface of Injections Evaluable Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the skin surface of injections. Only participants with a positive surface of injection site qPCR test were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 16 | 3 | 18 | 16 | 6 | 11 | 8 | 4 | 6
percentage of participants | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 20.6] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 28.5] | 12.5 [0.3 to 52.7] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 45.9]

18. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA at the Exterior of the Occlusive Dressing
Description: The percentage of participants with positive qPCR and subsequent positive plaque assays were evaluated from swabs of the exterior of the occlusive dressing. Detectable DNA was defined as a positive result by qPCR analysis.
Time Frame: Week 1 to Week 7
Population: Exterior of Occlusive Dressing Evaluable Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the exterior of the occlusive dressing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 23 | 21 | 9 | 12 | 9 | 5 | 7
percentage of participants | 30.4 [13.2 to 52.9] | 20.0 [0.5 to 71.6] | 39.1 [19.7 to 61.5] | 61.9 [38.4 to 81.9] | 66.7 [29.9 to 92.5] | 33.3 [9.9 to 65.1] | 44.4 [13.7 to 78.8] | 60.0 [14.7 to 94.7] | 14.3 [0.4 to 57.9]

19. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus at the Exterior of the Occlusive Dressing
Description: The percentage of participants with detectable virus were evaluated from swabs of the exterior of the occlusive dressings. Detectable virus was defined as a positive result by TCID50.
Time Frame: Week 1 to Week 7
Population: Exterior of Occlusive Dressing Evaluable Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the exterior of the occlusive dressing. Only participants with a positive exterior of occlusive dressing qPCR test were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 7 | 1 | 9 | 13 | 6 | 4 | 4 | 3 | 1
percentage of participants | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 24.7] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5]

20. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA at the Oral Mucosa
Description: The percentage of participants with positive qPCR and subsequent positive plaque assays were evaluated from swabs of the oral mucosa. Detectable DNA was defined as a positive result by qPCR analysis.
Time Frame: Part 1: Week 1 to Week 37. Part 2: Week 1 to Week 43
Population: Oral Mucosa Evaluable Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the oral mucosa.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 23 | 5 | 24 | 22 | 10 | 16 | 10 | 5 | 10
percentage of participants | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 52.2] | 29.2 [12.6 to 51.1] | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 30.8] | 12.5 [1.6 to 38.3] | 10.0 [0.3 to 44.5] | 60.0 [14.7 to 94.7] | 10.0 [0.3 to 44.5]

21. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus at the Oral Mucosa
Description: The percentage of participants with detectable virus were evaluated from swabs of the oral mucosa. Detectable virus was defined as a positive result by TCID50.
Time Frame: Week 1 to Week 7
Population: Oral Mucosa Evaluable Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the oral mucosa. Only participants with a positive oral mucosa qPCR test were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 0 | 0 | 7 | 1 | 0 | 2 | 1 | 3 | 1
percentage of participants |  |  | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 97.5] |  | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5]

22. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA in Lesions Suspected to be Herpetic in Origin
Description: The percentage of participants with positive qPCR were evaluated in any swab of a lesion suspected to be herpetic in origin. Detectable DNA was defined as a positive result by qPCR analysis.
  Participants returned to the clinic within 3 days of the occurrence of reportable lesion suspected to be herpetic in origin such as cold sores or vesicles. The lesion was evaluated by the Investigator and swabbed if herpes simplex virus infection was suspected.
Time Frame: Day 1 to 30 days post-last dose of talimogene laherparepvec. The maximum duration of talimogene laherparepvec treatment was 102.4 weeks and pembrolizumab treatment was 109.3 weeks.
Population: Reactive Swab Analysis Set: Included participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab sample collected from lesions that were suspected to be herpetic in origin.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
Number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
percentage of participants | 0.0 [0.0 to 84.2] |  |  | 100.0 [2.5 to 100.0] |  |  |  |  |

ADVERSE EVENTS:
Time Frame: From the first dose date to the earlier of 90 days for treatment-emergent SAEs or 30 days for other (non-serious) TEAEs after the last dose date (talimogene laherparepvec or pembrolizumab, whichever is later) or the participants initiate new therapy. Median [min, max] duration of exposure was 6.1 [0.1, 33.1] weeks in Part 1 monotherapy cohorts, 9.2 [0.1, 98.3] weeks in Part 1 combination cohorts and 6.1 [0.1, 109.3] weeks in Part 2. All-cause mortality was reported from Day 1 to up to 297 weeks.
Arm/Group | Part 1: Monotherapy Group A | Part 1: Monotherapy Group B | Part 1: Combination Therapy Group A | Part 1: Combination Therapy Group B | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) | Part 2: Triple Negative Breast Cancer (TNBC) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) | Part 2: Basal Cell Carcinoma (BCC) | Part 2: Colorectal Adenocarcinoma (CRC)
All-Cause Mortality (participants affected / at risk) | 21/23 | 3/5 | 22/24 | 14/22 | 8/10 | 13/18 | 5/10 | 4/5 | 8/10
Serious Adverse Events (participants affected / at risk) | 10/23 | 2/5 | 10/24 | 11/22 | 4/10 | 7/18 | 5/10 | 3/5 | 3/10
Other Adverse Events (participants affected / at risk) | 23/23 | 5/5 | 24/24 | 21/22 | 10/10 | 15/18 | 8/10 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Monotherapy Group A (N=23) | Part 1: Monotherapy Group B (N=5) | Part 1: Combination Therapy Group A (N=24) | Part 1: Combination Therapy Group B (N=22) | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) (N=10) | Part 2: Triple Negative Breast Cancer (TNBC) (N=18) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) (N=10) | Part 2: Basal Cell Carcinoma (BCC) (N=5) | Part 2: Colorectal Adenocarcinoma (CRC) (N=10)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 4 | 1 | 2 | 2 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Monotherapy Group A (N=23) | Part 1: Monotherapy Group B (N=5) | Part 1: Combination Therapy Group A (N=24) | Part 1: Combination Therapy Group B (N=22) | Part 2: Hormone Receptor Positive Breast Cancer (HRBC) (N=10) | Part 2: Triple Negative Breast Cancer (TNBC) (N=18) | Part 2: Cutaneous Squamous Cell Carcinoma (CSCC) (N=10) | Part 2: Basal Cell Carcinoma (BCC) (N=5) | Part 2: Colorectal Adenocarcinoma (CRC) (N=10)
Anaemia (Blood and lymphatic system disorders) | 7 | 0 | 6 | 3 | 2 | 3 | 1 | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 6 | 8 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 6 | 1 | 3 | 0 | 1 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 0 | 4 | 1 | 3 | 0 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 5 | 2 | 4 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 14 | 4 | 7 | 3 | 2 | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 2 | 8 | 5 | 5 | 3 | 1 | 0 | 2
Application site pain (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 5 | 2 | 3 | 5 | 0 | 0 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 4 | 1 | 13 | 8 | 8 | 0 | 2 | 0 | 3
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 11 | 1 | 8 | 4 | 3 | 1 | 1 | 2 | 5
Influenza like illness (General disorders) | 2 | 0 | 2 | 3 | 1 | 1 | 2 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 3 | 4 | 2 | 1 | 2 | 0 | 4
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 18 | 4 | 22 | 17 | 9 | 8 | 3 | 1 | 9
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver tenderness (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated adverse reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex viraemia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 1 | 3 | 0 | 3 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 6 | 2 | 2 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 3 | 0 | 3 | 2 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Blood creatinine abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
CD4 lymphocyte percentage decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Creatinine renal clearance increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroxine free decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0 | 5 | 2 | 3 | 1 | 0 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4 | 3 | 2 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5 | 1 | 1 | 1 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 2 | 6 | 2 | 4 | 1 | 0 | 0 | 0
Hypergeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 1 | 3 | 2 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 6 | 6 | 0 | 2 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 2 | 1 | 1 | 3 | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mass excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 6 | 2 | 1 | 2 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT02509507/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT02509507/SAP_001.pdf